CLINICAL TRIAL: NCT00089908
Title: Phase I Study of the Safety and Immunogenicity of rDEN1delta30, a Live Attenuated Virus Vaccine Candidate for the Prevention of Dengue Serotype 1
Brief Title: Safety of and Immune Response to a Dengue Virus Vaccine (rDEN1delta30) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Anna Durbin, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 199; H.22.04.04.23.B2
Record Dates: First submitted 2004-08-17; First posted 2004-08-19 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Dengue Fever
Keywords: Dengue Vaccine; Dengue Virus; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): One subcutaneous vaccination with rDEN1delta30 vaccine (10^3 PFU dose) into the deltoid region of either arm.
  Interventions: Biological: rDEN1delta30
- 2 (Experimental): One subcutaneous vaccination with rDEN1delta30 vaccine (10^5 PFU dose) into the deltoid region of either arm. This arm may enroll after Arm 1 depending on the effect of the vaccine on subjects in Arm 1.
  Interventions: Biological: rDEN1delta30
- 3 (Placebo Comparator): One subcutaneous vaccination with placebo into the deltoid region of either arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rDEN1delta30 — Live attenuated rDEN1delta30 vaccine
  Arms: 1; 2
Biological: Placebo — Placebo for rDEN1delta30
  Arms: 3

SUMMARY:
Dengue fever, which is caused by dengue viruses, is a major health problem in tropical and subtropical regions of the world. The purpose of this study is to test the safety of and immune response to a new dengue virus vaccine in healthy adults.

DETAILED DESCRIPTION:
More than 2 billion people living in tropical and subtropical regions of the world are at risk of dengue virus infection. Dengue viruses cause dengue fever, as well as the more severe dengue hemorrhagic fever/shock syndrome, and dengue virus infection is the leading cause of hospitalization and death in children in several tropical Asian countries. This study will evaluate the safety and immunogenicity of a live, attenuated dengue virus called rDEN1delta30, which is derived from the Western Pacific DEN1 serotype.

This study will last 180 days. Participants in Cohort 1 will be randomly assigned to receive rDEN1delta30 or placebo at study entry. Cohort 2 will begin only after safety review of all participants in Cohort 1. Participants in Cohort 2 will receive a higher dose of rDEN1delta30 or placebo.

After vaccination, participants will be asked to monitor their temperature every day for 16 days. Study visits will occur every other day after vaccination until Day 16, followed by 4 additional visits at selected days through Day 180. Blood collection and a targeted physical exam will occur at each study visit. Some participants will be asked to undergo a skin biopsy or additional blood collection at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Willing to be followed for the duration of the study
* Willing to use acceptable methods of contraception
* Good general health

Exclusion Criteria:

* Clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the volunteer to understand and cooperate with the study
* Liver, renal, or hematologic disease
* Alcohol or drug abuse within 12 months of study entry
* History of severe allergic reaction or anaphylaxis
* Emergency room visit or hospitalization for severe asthma within 6 months of study entry
* HIV-1 infected
* HCV infected
* Hepatitis B surface antigen positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days of study entry. Participants who have used topical or nasal corticosteroids are not excluded.
* Live vaccine within 4 weeks of study entry
* Killed vaccine within 2 weeks of study entry
* Blood products within 6 months of study entry
* Investigational drugs or vaccines within 60 days prior to study entry or while currently enrolled in this clinical trial
* Previously received a licensed or experimental yellow fever or dengue vaccine
* Surgical removal of spleen
* History of dengue virus infection or other flavivirus infection
* Other condition that, in the opinion of the investigator, would affect the participant's participation in the study
* Pregnancy or breastfeeding
* Plan to travel to an area where dengue infection is common

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Determine the frequency of vaccine related AEs for each dose graded by severity | Throughout study
Determine the amount of dengue 1 neutralizing antibody induced by the vaccine | At Day 42

SECONDARY OUTCOMES:
To assess the durability of the antibody response | At Day 180
To assess the frequency, quantity, and duration of viremia in each dose cohort studied | Throughout study
To compare the T cell mediated immune response against dengue viruses of those volunteers infected with the rDEN1delta30 vaccine virus with that of uninfected volunteers and placebo recipients | Throughout study
If both doses of vaccine are administered, to compare the infectivity rates, safety, and immunogenicity between dose groups | At study completion
To evaluate the immunopathological mechanism of vaccine-associated rash in those volunteers who are willing to undergo skin biopsy | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research, John Hopkins School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Jacobs M, Young P. Dengue vaccines: preparing to roll back dengue. Curr Opin Investig Drugs. 2003 Feb;4(2):168-71. PMID 12669377
- [Background] Pang T. Vaccines for the prevention of neglected diseases--dengue fever. Curr Opin Biotechnol. 2003 Jun;14(3):332-6. doi: 10.1016/s0958-1669(03)00061-2. PMID 12849789
- [Background] Rothman AL. Dengue: defining protective versus pathologic immunity. J Clin Invest. 2004 Apr;113(7):946-51. doi: 10.1172/JCI21512. PMID 15057297
- [Background] Sun W, Edelman R, Kanesa-Thasan N, Eckels KH, Putnak JR, King AD, Houng HS, Tang D, Scherer JM, Hoke CH Jr, Innis BL. Vaccination of human volunteers with monovalent and tetravalent live-attenuated dengue vaccine candidates. Am J Trop Med Hyg. 2003 Dec;69(6 Suppl):24-31. doi: 10.4269/ajtmh.2003.69.6_suppl.0690024. PMID 14740952